CLINICAL TRIAL: NCT06048354
Title: Double Blind, Randomized, Placebo Controlled Clinical and Instrumental Evaluation of the Efficacy of Two Dietary Supplements Claiming Anti-aging Properties
Brief Title: Evaluation of the Efficacy of Two Dietary Supplements Claiming Anti-aging Properties
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seppic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IT0003398/21
Record Dates: First submitted 2023-08-31; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Wheat Polar Lipid Complex Oil (Experimental): Dietary supplement - Wheat Polar Lipid Complex (Oil)
  Interventions: Dietary Supplement: Wheat Polar Lipid Complex Oil
- Wheat Polar Lipid Complex Powder (Experimental): Dietary supplement - Wheat Polar Lipid Complex (Powder)
  Interventions: Dietary Supplement: Wheat Polar Lipid Complex Powder
- Placebo (Placebo Comparator): Dietary supplement - Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Wheat Polar Lipid Complex Oil — The study foresees the intake of 2 capsules per day during 84 days
  Arms: Wheat Polar Lipid Complex Oil
Dietary Supplement: Wheat Polar Lipid Complex Powder — The study foresees the intake of 2 capsules per day during 84 days
  Arms: Wheat Polar Lipid Complex Powder
Dietary Supplement: Placebo — The study foresees the intake of 2 capsules per day during 84 days
  Arms: Placebo

SUMMARY:
The study is aimed to assess the efficacy of two dietary supplements composed of a Wheat Polar Lipid Complex (WPLC) in reducing skin aging signs, in particular in improving firmness/elasticity, skin moisturization and skin surface properties.

DETAILED DESCRIPTION:
A double blind, parallel groups, placebo-controlled study is carried out on 72 healthy female subjects aged between 30 and 60 years old showing slight-moderate clinical signs of skin aging over the face. The study foresees 56 days of products intake. Evaluations of the parameters under study are performed at baseline, after 14, 28 and 56 days of products consumption. Moreover post-treatment evaluations are performed 56 days after the end of product intake.

ELIGIBILITY:
Inclusion criteria :

* Healthy female subjects,
* Caucasian ethnicity,
* Age between 30 and 60 years old (extremes included),
* Wrinkles related to chronological ageing (from mild to moderate),
* Wrinkles related to photo-ageing (medium photo-ageing signs, dry and devitalized skin, asphyxia, pale and greyish skin, early ageing signs caused by a slowing in the cells activity),
* Subjects with dry skin defined with corneometric index < 50 a.u.,
* Body mass index BMI between 19 and 30,
* At least 10 menopause women per group,
* Subjects who have not been recently involved in any other similar study (evaluation is performed case by case by the experimenter but at least 1 month must be elapsed between a previous study on food supplement),
* Willingness not to use chemical products or treatments on hair and nails (such as hair colour, straightening, permanent nail polish) in the two weeks preceding T56 visit,
* Willingness to not use during the study period products other than the test product,
* Willingness to not vary the normal diet and daily routine (at the beginning of the study volunteers list their usual routine: sport activities, sleeping habits, etc. ),
* Subjects under effective contraception (oral/not oral) if women of childbearing potential; not expected to be changed during the trial,
* Subjects who have not sun exposure (both natural or artificial) for at least two months
* Subjects who accept not to expose in intensive way to UV rays during the whole study duration,
* Willingness not to use similar products that could interfere with the product to be tested,
* Subject aware of the study procedures and having signed an informed consent form.

Exclusion Criteria:

* Subject does not meet the inclusion criteria,
* Subject with known or suspected sensitization to one or more test formulation ingredients,
* Any condition that the principal investigator deems inappropriate for participation,
* Pregnant/breastfeeding female or who have planned a pregnancy during the study period,
* Pharmacological treatments (topic or systemic) known to interfere with skin metabolism/physiology,
* Lipid metabolism disorders (hypercholesterolemia, hyperlipidemia) and following treatment for theses disease,
* Subjects under locally pharmacological treatment on the skin area monitored during the test,
* Subjects under treatment with food supplements which could interfere with the functionality of the product under study,
* Subjects which show skin alterations on the monitored area which could interfere with the functionality of the product under study,
* Subjects who underwent to botox, hyaluronic acid, collagen injections or each type of facial surgery in the past 6 months,
* Severe concurrent diseases,
* Adult protected by the law (under guardianship, or hospitalized in a public or private institution, for a reason other than the research, or incarcerated),
* Subject is unable to communicate or cooperate with the Investigator due to language problems, poor mental development, or impaired cerebral function,
* Subjects resulting positive to Sars-Cov. 19 in the past 6 months/ during the study
* Subjects not presenting a valid Greenpass.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Skin moisturization | Baseline
  Skin moisturization is measured by the Corneometer®, which analyze the dielectric constant and therefore the water content of the skin
Skin moisturization | 14 days
  Skin moisturization is measured by the Corneometer®, which analyze the dielectric constant and therefore the water content of the skin
Skin moisturization | 28 days
  Skin moisturization is measured by the Corneometer®, which analyze the dielectric constant and therefore the water content of the skin
Skin moisturization | 56 days
  Skin moisturization is measured by the Corneometer®, which analyze the dielectric constant and therefore the water content of the skin
Skin moisturization | 56 days post supplementation
  Skin moisturization is measured by the Corneometer®, which analyze the dielectric constant and therefore the water content of the skin

SECONDARY OUTCOMES:
Skin elasticity | Baseline
  Skin elasticity measurement is based on the suction/elongation method and the subsequent release of the skin inside the opening of the instrument (Cutometer®)
Skin elasticity | 14 days
  Skin elasticity measurement is based on the suction/elongation method and the subsequent release of the skin inside the opening of the instrument (Cutometer®)
Skin elasticity | 28 days
  Skin elasticity measurement is based on the suction/elongation method and the subsequent release of the skin inside the opening of the instrument (Cutometer®)
Skin elasticity | 56 days
  Skin elasticity measurement is based on the suction/elongation method and the subsequent release of the skin inside the opening of the instrument (Cutometer®)
Skin elasticity | 56 days post supplementation
  Skin elasticity measurement is based on the suction/elongation method and the subsequent release of the skin inside the opening of the instrument (Cutometer®)
Transepidermal water loss | Baseline
  The water evaporating from the skin is measured using a probe (Tewameter®) that detect changes in water vapor density
Transepidermal water loss | 14 days
  The water evaporating from the skin is measured using a probe (Tewameter®) that detect changes in water vapor density
Transepidermal water loss | 28 days
  The water evaporating from the skin is measured using a probe (Tewameter®) that detect changes in water vapor density
Transepidermal water loss | 56 days
  The water evaporating from the skin is measured using a probe (Tewameter®) that detect changes in water vapor density
Transepidermal water loss | 56 days post supplementation
  The water evaporating from the skin is measured using a probe (Tewameter®) that detect changes in water vapor density
Skin roughness | Baseline
  Skin roughness (Rz parameter) is measured by Primos CR, a 3D scanner using fringe projection to measure skin surface properties
Skin roughness | 14 days
  Skin roughness (Rz parameter) is measured by Primos CR, a 3D scanner using fringe projection to measure skin surface properties
Skin roughness | 28 days
  Skin roughness (Rz parameter) is measured by Primos CR, a 3D scanner using fringe projection to measure skin surface properties
Skin roughness | 56 days
  Skin roughness (Rz parameter) is measured by Primos CR, a 3D scanner using fringe projection to measure skin surface properties
Skin roughness | 56 days post supplementation
  Skin roughness (Rz parameter) is measured by Primos CR, a 3D scanner using fringe projection to measure skin surface properties
Skin smoothness | Baseline
  Skin smoothness (Ra parameter) is measured by Primos CR, a 3D scanner using fringe projection to measure skin surface properties
Skin smoothness | 14 days
  Skin smoothness (Ra parameter) is measured by Primos CR, a 3D scanner using fringe projection to measure skin surface properties
Skin smoothness | 28 days
  Skin smoothness (Ra parameter) is measured by Primos CR, a 3D scanner using fringe projection to measure skin surface properties
Skin smoothness | 56 days
  Skin smoothness (Ra parameter) is measured by Primos CR, a 3D scanner using fringe projection to measure skin surface properties
Skin smoothness | 56 days post supplementation
  Skin smoothness (Ra parameter) is measured by Primos CR, a 3D scanner using fringe projection to measure skin surface properties
Wrinkle depth | Baseline
  Wrinkle depth (Sv parameter) is measured by Primos CR, a 3D scanner using fringe projection to measure skin surface properties
Wrinkle depth | 14 days
  Wrinkle depth (Sv parameter) is measured by Primos CR, a 3D scanner using fringe projection to measure skin surface properties
Wrinkle depth | 28 days
  Wrinkle depth (Sv parameter) is measured by Primos CR, a 3D scanner using fringe projection to measure skin surface properties
Wrinkle depth | 56 days
  Wrinkle depth (Sv parameter) is measured by Primos CR, a 3D scanner using fringe projection to measure skin surface properties
Wrinkle depth | 56 days post supplementation
  Wrinkle depth (Sv parameter) is measured by Primos CR, a 3D scanner using fringe projection to measure skin surface properties
Self-assessment of product efficacy | 56 days
  Questionnaire (20 questions with 4 possible answers : completely agree / agree / disagree / completely disagree)
Skin lipidic profile | Baseline
  Untargeted lipidomic analysis : Extraction of lipids from skin stripping and quantification by ultra-high performance liquid chromatography coupled to mass spectrometry (relative peak intensity)
Skin lipidic profile | 56 days
  Untargeted lipidomic analysis : Extraction of lipids from skin stripping and quantification by ultra-high performance liquid chromatography coupled to mass spectrometry (relative peak intensity)

CONTACTS AND LOCATIONS:
Overall Officials: Ileana De Ponti, Study Director — Complife Italia S.r.l
Locations (1):
- Complife Italia srl, Milan, Italy